CLINICAL TRIAL: NCT06136312
Title: A Clinical Investigation to Confirm Performance and Safety of the Multi4 System in Patients With Suspected Recurrent Bladder Cancer Lesions
Brief Title: Clinical Investigation of the Multi4 System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Multi4 Medical Ab (Industry)
Collaborators: Key2Compliance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-02-23-0002
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Multi4 procedure (Experimental): Complete TURBT procedure performed in local anesthesia with Multi4 instrument via flexible cystoscopy
  Interventions: Device: Multi4

INTERVENTIONS:
Device: Multi4 — TURBT procedure performed with the Multi4 instrument in local anesthesia

SUMMARY:
A Clinical Investigation to Confirm Performance and Safety of the Multi4 System in Patients with Suspected Recurrent Bladder Cancer Lesions

DETAILED DESCRIPTION:
The overall purpose of this study is to confirm performance and safety of Multi4 Medical Device System when used as intended: to cauterize, remove, and automatically collect multiple tissue samples through the working channel of an endoscope.

The safety profile will be documented by collecting data on frequency and severity of complications, AEs such as bleeding and perforations.

ELIGIBILITY:
Inclusion Criteria:

* Previous bladder cancer Ta/T1 G1-3
* Recurrence of urinary superficial/ non-muscle-invasive bladder cancer visible at cystoscopy, estimated size < 10 mm
* Willingness and ability to provide informed consent
* Age ≥18 years

Exclusion Criteria:

* Implantable Cardioverter Defibrillator (ICD) that cannot be inactivated
* Current/ongoing untreated urinary tract infection
* Pregnancy or breastfeeding
* Be identified by the Investigator as inappropriate from a medical or compliance perspective to participate in this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Evaluable biopsies | At procedure
  Biopsies collected by the instrument are evaluable by pathologist

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | One week
  Frequency and severity of adverse events related to instrument use
Number of patients with complete procedures performed | At procedure
  Proportion of procedures that can be completely performed with the instrument
Patient-reported treatment-related pain (numeric rating scale) | At procedure
  Patient reported pain experienced during procedure, from 0 (no pain) to 10 (worst possible pain)
Quality of life (EQ-5D-5L) | At procedure and after 1 week
  Difference in self reported quality of life with the EuroQol 5-level instrument, prior to procedure compared to one week after procedure
Time to perform procedure | At procedure
  Time taken to perform a complete procedure
Time for patient surveillance | At procedure
  Time taken for observation after procedure
Self reported satisfaction with procedure | One week
  Proportion of patients who, in case of further bladder cancer recurrences, would choose to undergo the same procedure in local anesthesia as opposed to a full TURBT in general anesthesia
Operator-reported ease of use | At procedure
  Number of procedures where to operator reports that the Multi4 instrument works without issue and is easily handled (yes), or whether there are handling issues (no)
Cost effectiveness | At procedure
  Total costs associated with procedure compared to a complete TURBT in general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kjölhede, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No